CLINICAL TRIAL: NCT00626834
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Intravenous Cocaine and Oral Gamma Vinyl-Gamma-Amino Butyric Acid (VIGABATRIN) Interaction Study
Brief Title: Vigabatrin Ph 1 Cocaine Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OV-1014
Record Dates: First submitted 2008-02-18; First posted 2008-02-29 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-08

CONDITIONS: Cocaine Addiction
Keywords: cocaine addiction; vigabatrin; ovation pharmaceuticals; cocaine; cocaine related disorders; behavior addictive; mental disorders; therapeutic uses; physiologic effects of drugs; disorder of environmental origin; central nervous system stimulants; central nervous system agents; pharmacological actions; substance related disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive; Mental Disorders; Substance-Related Disorders | interventions — Vigabatrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vigabatrin Dose 1 (Experimental)
  Interventions: Drug: Vigabatrin
- Vigabatrin Dose 2 (Experimental)
  Interventions: Drug: Vigabatrin
- Vigabatrin Dose 3 (Experimental)
  Interventions: Drug: Vigabatrin
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Vigabatrin — Dose 1 BID
  Arms: Vigabatrin Dose 1
Drug: Vigabatrin — Dose 2 BID
  Arms: Vigabatrin Dose 2
Drug: Vigabatrin — Dose 3 BID
  Arms: Vigabatrin Dose 3
Drug: Matching placebo — Matching placebo BID
  Arms: Matching placebo

SUMMARY:
This is a Phase 1 safety/tolerably study to determine if there are clinically significant interactions between oral vigabatrin (gamma vinyl-gamma-amino butyric acid; VGB) concurrent with intravenous (IV) cocaine infusions.

DETAILED DESCRIPTION:
STUDY DESIGN: This is a randomized, double-blind, placebo-controlled, parallel group study of the effects of VGB compared to placebo control on the physiological and subjective effects of IV infusions of cocaine (cocaine experienced volunteers).

Subjects will be randomized within each clinical site to one of four groups (placebo control or one of three doses of VGB twice daily).During VGB steady state dosing, subjects will receive double-blind infusions of saline and cocaine. Subjects will be asked to return for follow-up approximately 7 and 14 days after the day of clinic discharge.

STUDY DURATION: The maximum duration is 56 days, including 14 inpatient days of assessments and investigational products administration, and two follow-up visits after clinic discharge.

SAMPLE SIZE: Twenty-four subjects will be randomized to one of three doses of vigabatrin or placebo.

POPULATION: Volunteer, cocaine-experienced, non-treatment seeking cocaine users, 18 to 45 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 45 years of age, inclusive
* Currently be a non-treatment seeking cocaine user as confirmed by a positive urine test for cocaine
* Able to provide written informed consent
* A negative pregnancy test within 72 hours prior to receiving the first infusion of cocaine

Exclusion Criteria:

Please contact site for more information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
safety/tolerability and AE assessments including HR/BP/ECG/QTc | 56 days

SECONDARY OUTCOMES:
VGB/PK during cocaine infusions and effect of VGB on cocaine craving | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John D. Roache, Ph.D., Principal Investigator — University of Texas; Nora Chiang, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA); Ahmed Elkashef, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA); Roberta Kahn, M.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No